CLINICAL TRIAL: NCT02196545
Title: An Easily Accessible Physical Activity Training Program for Patients With Alzheimer's Dementia: Effect on Clinical and Neurobiological Parameters (MOTODEM)
Brief Title: Physical Activity Training Program for Patients With Alzheimer's Dementia
Acronym: MOTODEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: RECK-Technik GmbH & Co. KG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTDEM-001
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Exercise, patients train on a specifically programmed movement trainer three times a week for 30 minutes (total duration 12 weeks)
  Interventions: Behavioral: Exercise
- Treatment as usual (No Intervention): Treatment according to guidelines of German Society for Psychiatry, Psychotherapy and Nervous Diseases (DGPPN) and German Society of Neurology (DGN) without movement trainer exercise

INTERVENTIONS:
Behavioral: Exercise
  Other Names: (RECK MotoMed®)
  Arms: Exercise

SUMMARY:
The purpose of this study is to determine if a home based physical activity training program for patients with Alzheimer's dementia has effects on clinical and neurobiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* age >55 years
* German is the dominant language (necessary for neuropsychological testing)
* minimum of 8 years formal school education
* caregiver (e.g. spouse) living at home with participant
* physical examination does not reveal contraindications to physical activity
* stable dose of pharmacological dementia treatment according to German guidelines (DGPPN) with acetylcholinesterase inhibitor or memantin or combination for at least 6 months
* no other medication that could influence cognitive functioning (e.g. benzodiazepines, sleep aids, neuroleptics)

Exclusion Criteria:

* history of neurological or psychiatric disease other than AD
* history of substance abuse disorder
* history of electroconvulsive therapy (ECT) during the last 6 months
* structural brain deficits diagnosed in the MRI scan, also without clinical relevance (incidental finding)
* pacemaker, artificial heart valve, insulin pump or other medical implants
* average steps/day are above 10.000 steps/day

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
activities of daily living | change from baseline after 12 weeks
  Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS/ADL)

SECONDARY OUTCOMES:
behavioral symptoms of dementia | change from baseline after 12 weeks and 24 weeks
  Neuropsychiatric Inventory (NPI) total score
cognition | change from baseline after 12 weeks and 24 weeks
  Mini Mental Status Examination (MMSE)
executive function and language ability | change from baseline after 12 weeks and 24 weeks
  semantic and phonemic word fluency
caregiver burden | change from baseline after 12 weeks and 24 weeks
  Neuropsychiatric inventory (NPI) total burden score
Reaction time, hand-eye quickness and attention | change from baseline after 12 weeks and 24 weeks
  Ruler Drop Test
activities of daily living | change from baseline after 24 weeks
  Alzheimer's Disease Cooperative Study/Activities of Daily Living (ADCS/ADL)

OTHER OUTCOMES:
hippocampal cortical thickness | change from baseline after 12 weeks
  subregional hippocampal cortical thickness based on MRI analyses

CONTACTS AND LOCATIONS:
Overall Officials: Vjera A Holthoff, Prof., Principal Investigator — Technische Universität Dresden
Locations (1):
- Technische Universität Dresden, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Holthoff VA, Marschner K, Scharf M, Steding J, Meyer S, Koch R, Donix M. Effects of physical activity training in patients with Alzheimer's dementia: results of a pilot RCT study. PLoS One. 2015 Apr 17;10(4):e0121478. doi: 10.1371/journal.pone.0121478. eCollection 2015. PMID 25884637